CLINICAL TRIAL: NCT06179121
Title: "Adding DNA-test for Screening of HLA-DQ2 and DQ8 to Improve the Early Diagnosis of Celiac Disease at the Dutch Preventive Youth Healthcare Centres (GLUTEN-GEN)"
Brief Title: "Adding DNA-test for Screening of HLA-DQ2 and DQ8 to Improve Early Diagnosis of Celiac Disease"
Acronym: GLUTEN-GEN
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, crmeijerboekel, PhD, Leiden University Medical Center
Other Study IDs: P23.025 (METC LDD); 05550402110016 (Other Grant/Funding Number: ZonMw ("Preventie Vroege opsporing" program))
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Celiac Disease in Children
Keywords: Coeliac disease; Preventive Youth Health Care Center
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA acquired from dried blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1 Cohort (Validation of HLA- DQ2/8 typing): Children (1-18 years old) coming for consultation at the LUMC for (suspicion of) CD
  Interventions: Other: DNA test for screening HLA-DQ2 and DQ8 from dried blood spots to early detect Celiac Disease
- Phase 2 Cohort (Implementation of HLA-DQ2/8 typing on the Preventive YHCCs): Children (12 months to 4 years old), at least with one of the 10 CD-related symptoms, not diagnosed with CD, and not on a GFD,
  Interventions: Other: DNA test for screening HLA-DQ2 and DQ8 from dried blood spots to early detect Celiac Disease

INTERVENTIONS:
Other: DNA test for screening HLA-DQ2 and DQ8 from dried blood spots to early detect Celiac Disease — Phase 1 and 2: After blood collection (in combination with regular care) and informed consent, a blood droplet obtained by an additional fingerprick (Phase 1 and just an extra droplet from an existing finger prick for Phase 2) will be deposited on filter paper S&S 903™ (Schleicher and Schuell). DNA will be isolated using the QIAamp method designated for this purpose from dried blood spots (Qiagen). The results of the HLA-DQ2 and DQ8-typing using the dried blood spots will be compared with the results of the traditional HLA-typing. Factors that may influence the quality of the material will be taken into account in the validation process.

SUMMARY:
Celiac Disease (CD) is an immune-mediated systemic disorder elicited by the ingestion of gluten containing cereals from the normal diet, among others wheat, rye and barley. The disease is characterized by a variable combination of gluten-dependent clinical manifestations, CD specific antibodies, human leukocyte antigen (HLA)-DQ2 or HLA-DQ8 haplotypes and chronic inflammation of the small bowel.CD is one of the most common lifelong food- related disorders; it has a frequency of 1% in the general population: this corresponds to 170.000 persons in the Netherlands, and of them at least 30.000 children. However, CD is frequently unrecognized, partially because of its variable clinical presentations and symptoms. That timely diagnosis and treatment of CD could be achieved by active case-finding, show the preliminary results of the ongoing ZonMw sponsored project GLUTENSCREEN (531002001; www.glutenscreen.nl). Currently, HLA-typing is not a part of GLUTENSCREEN because current technique presents important drawbacks in settings without the availability of a laboratory. We here propose to develop a novel test for DNA isolation for HLA typing extracted from the dried blood spots obtained from the POCT at the Preventive YHCCs for early detection of CD. Repeated testing for CD could be omitted in children tested HLA-DQ2/8 negative, this reflects to 60% of the targeted population. To embed this technique in the case finding setting at the YHCCs, the test will be offered to a significant part of the general Dutch population between 0-4 years old, since more than 95% of the general population visit the YHCC. Primary Objective: To validate the HLA-DQ typing in blood taken by a fingerprick; to make it feasible in the regular Preventive YHCCs organization. Study population: Phase 1: From 50 children attending the LUMC dept. of Pediatrics because of suspected CD in whom traditional HLA-typing is part of their standard of care or from children with diagnosed CD in whom their HLA typing is already known. Phase 2: All parents of symptomatic children, 1-4 years of age, who visit the Preventive YHCC in the region of Kennemerland, will be asked to participate in this study.

DETAILED DESCRIPTION:
Celiac Disease (CD) is an immune-mediated systemic disorder elicited by the ingestion of gluten containing cereals from the normal diet, among others wheat, rye and barley. The disease is characterized by a variable combination of gluten-dependent clinical manifestations, CD specific antibodies, human leukocyte antigen (HLA)-DQ2 or HLA-DQ8 haplotypes and chronic inflammation of the small bowel[1,2]. T-cells in the lamina propria of the small bowel recognize the gluten peptides when they are bound to the HLA class II specificities DQ2 and/or DQ8 on antigen-presenting cells.

CD is one of the most common lifelong food- related disorders; it has a frequency of 1% in the general population: this corresponds to 170.000 persons in the Netherlands, and of them at least 30.000 children[3-7]. However, CD is frequently unrecognized, partially because of its variable clinical presentations and symptoms, ranging from malabsorption with chronic diarrhoea, poor growth in children and weight loss, to nonspecific signs and symptoms like chronic fatigue, osteoporosis/reduced bone mineral density, gastrointestinal symptoms or elevated liver enzymes [5,7,8]. Unrecognized and thereby undiagnosed and untreated disease is associated with short- and long-term complications such as delayed puberty, neuropsychiatric disturbances, associated autoimmune disease, miscarriages, small-for-date-births, osteoporosis, and, rarely, malignancy. CD has a considerable health burden for society and yields extensive negative economic consequences, thereby presenting a resource challenge for current and future health systems [9]. Once diagnosed, the patient's health status improves after treatment with a gluten free diet (GFD).

That timely diagnosis and treatment of CD could be achieved by active case-finding, show the preliminary results of the ongoing ZonMw sponsored project GLUTENSCREEN (531002001; www.glutenscreen.nl). In this active case finding project, started at February 2019, all children aged 1-4 years who attend the Preventive Youth Health Care Centres (YHCCs) in the region of Kennemerland are yearly assessed for 10 CD-related symptoms during their regular consultation. If a child has one or more symptoms, the parents of the child are invited to participate. After informed consent, a point of care test (POCT) assessing CD-specific antibodies against tissue-transglutaminase (TGA) from a droplet of blood, is performed onsite at the YHCCs. If the POCT is positive (TGA present), CD is highly suspected and the child is referred to the Leiden University Medical Centre (LUMC) for diagnosis according to the standard of care[1,2]. The preliminary results of GLUTENSCREEN are beyond expectations: From the 14.917 children attending the YHCCs, 5.512 (37.0%) of them had one or more CD-related symptoms.

The parents of 3.203 (58.1%) children gave informed consent for a POC-test. In 61 (1.9%) children the POC-test was positive. After additional investigations at our hospital, CD was confirmed in 55 children (1.7% of the tested children) (serum IgA TGA >10xULN and IgA against endomysium (EMA) positive) and ruled out in 5 children with dubious/positive POC test: in two children HLA-DQ2/8 was negative with negative TGA in serum (ELISA-test), in 3 children with TGA <10 x ULN (ELISA-test) in whom small bowel biopsies showed Marsh 1 lesions. One child still needs to be seen in the hospital (parents refused till now) (www.glutenscreen.nl). From the parents who were invited for GLUTENSCREEN, almost 80% is willing to participate if the POCT could be performed during the regular visit at the YHCC. All health care professionals reported that early CD detection by case-finding adds value to the preventive care they offer at the YHCCs.

These preliminary results of our active CD case-finding project at the Preventive YHCCs in the Netherlands illustrate that early detection of CD at the Preventive YHC is feasible and well-accepted by parents and health care professionals.

In GLUTENSCREEN all symptomatic children will be annually tested for CD at the Preventive YHCCs till the age of 4 years. In the region Kennemerland, GLUTENSCREEN has already been implemented in the regular care and POCT will be performed during consultation. However, the development of CD requires genetic susceptibility, present in 40% of the general population. Since the disease almost exclusively occurs in individuals with the human leukocyte antigen (HLA)-DQ2 and/or HLA- DQ8 haplotypes, codified by chromosome 6. The absence of HLA-DQ2/-DQ8 can exclude the possibility or future development of CD with a certainty close to 100%. Because of the high negative predictive value of HLA-typing for development of CD, repeated CD testing will be unnecessary in HLA-DQ2/DQ8 negative individuals (60% of the general population) [10].

Currently, HLA-typing is not a part of GLUTENSCREEN because current technique presents important drawbacks in settings without the availability of a laboratory, like the Preventive Care setting as the YHCCs, since it requires DNA extraction. Material for DNA extraction is usually obtained from whole blood (minimum quantity 4-5 ml) or from other cells, such as buccal mucosa. However, venipunctures are not feasible at the YHCCs and buccal mucosa DNA extraction in children is time-consuming.

We here propose to validate and implement the test for DNA isolation for HLA typing extracted from the dried blood spots to early detection for CD on the Preventive YHCCs.

Other projects have shown that the usage of real-time polymerase chain reaction (RT-PCR) on DNA acquired from dried blood samples is successful and can easily be applied to HLA-DQ2/DQ8 typing in this setting[11].

Adding HLA-DQ2/8 typing to the case finding strategy for CD at the Preventive YHCC is innovative since HLA-typing for CD has not previously been done in dried blood spots in the proposed setting. Furthermore, embedding this technique represents a novel approach to active case-finding of CD and consequently will improve secondary prevention of CD by early diagnosis at the Preventive YHCCs.

The outcome of the proposed study will have impact on the active case finding procedure of CD at the YHCCs. Repeated testing for CD could be omitted in children tested HLA-DQ2/8 negative, this reflects to 60% of the targeted population. This study will result in:

1. More efficient and decrease of the burden of the HLA-DQ2/8 negative children: less children have to be tested.
2. Clarity of the acceptability of HLA typing for CD in parents from young children.
3. Costs saving by reducing unnecessary follow up of children. To embed this technique in the case finding setting at the YHCCs, the test will be offered to a significant part of the general Dutch population between 0-4 years old, since more than 95% of the general population visit the YHCC.

   * Consult references at the end of this document

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* age 1-18 years,
* consultation at the LUMC for (suspicion of) CD,
* parents have a sufficient knowledge of Dutch language,
* written informed consent from child and/or parent

Phase 2:

* age 12 months to 4 years,
* at least one of the 10 CD-related symptoms
* not diagnosed with CD,
* not on a GFD,
* parents have a sufficient knowledge of Dutch language,
* written informed consent from the parent(s)

Exclusion Criteria:

Phase 1 and 2:

* no informed consent,
* insufficient knowledge of Dutch language and/or inability to understand the information provided,
* bleeding disorders.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Phase 1: From 50 children attending the LUMC dept.of Pediatrics because of suspected CD in whom traditional HLA-typing is part of their standard of care or from children with diagnosed CD in whom their HLA typing is already known. The LUMC is a reference centre for CD in children. On the outpatient clinic, more than 90 children per 6 months will be seeing with (the suspicion) of CD and more than 500 children visit the clinic for the annual follow up of CD, which means that the number needed to validated the HLA-results are realistic.
  Phase 2 : All parents of symptomatic children, 1-4 years of age, who visit the Preventive YHCC in the region of Kennemerland, will be asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the HLA-test in dried blood spots will be calculated (Phase 1) | Month 6 to month 9 (total duration of the study: 18 months)
  The results of the HLA-DQ2 and DQ8-typing using the dried blood spots will be compared with the results of the traditional HLA-typing. DNA extraction for HLA-DQ typing from dry blood spots will be performed using the QIAamp method [12-15]. A protocol to isolate DNA has been developed and the isolation is executable by all the well skilled laboratory analysts. DNA extraction per sample takes about 15 minutes and it is possible to determine several samples at the same time. The equipment and optical technology are already present at the LUMC.
Prevalence of HLA-DQ2/8 in the general population (Phase 2) population (parents) and the health care professionals.(Phase 2) | Month 9 to month 12 (after the validation phase 1)
  Children with positive HLA-DQ2/8 typing (n/%), Children with negative HLA-DQ2/8 typing (n/%), Children in whom the test failed (including reason), Evaluation of the acceptance and impact of the HLA-typing for CD by the Dutchpopulation (parents) and the health care professionals For the HLA-DQ typing approximately 15 μL is necessary which corresponds with 1-2 droplets of blood. After informed consent, an extra droplet of blood will be collected for the novel HLA-DQ2/8 typing by the finger prick when performing the POCT for TGA determination as done in GLUTENSCREEN. The filter-papers will be stored, at room temperature, safely at the YHCCs. Once a week, all the collected filter papers with dried blood spots will be sent to the department of the Immunology in specially marked envelops. After the DNA isolation, HLA-DQ typing and interpretation.

SECONDARY OUTCOMES:
Cost-effectiveness of the investigational strategy (Time investment by medical and nursing staff at the YHCCs (sec), costs of the investigational strategy (time, materials) (€)) | Month 9 to month 12
  To evaluate the cost-effectiveness of case finding with and without HLA-DQ2/8 typing. This part of the study will be done by the health economist. Factors that will be included are cost for: the novel genetic test, health care professionals at the YHCC and laboratorial, storage and transport of the material for the genetic test. These costs will compared to the costs in the situation without HLA-DQ2/8 testing as done in GLUTENSCREEN

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Meijer-Boekel, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Centre (LUMC), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Husby S, Koletzko S, Korponay-Szabo IR, Mearin ML, Phillips A, Shamir R, Troncone R, Giersiepen K, Branski D, Catassi C, Lelgeman M, Maki M, Ribes-Koninckx C, Ventura A, Zimmer KP; ESPGHAN Working Group on Coeliac Disease Diagnosis; ESPGHAN Gastroenterology Committee; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. European Society for Pediatric Gastroenterology, Hepatology, and Nutrition guidelines for the diagnosis of coeliac disease. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):136-60. doi: 10.1097/MPG.0b013e31821a23d0. PMID 22197856
- [Result] Jansson-Knodell CL, Hujoel IA, West CP, Taneja V, Prokop LJ, Rubio-Tapia A, Murray JA. Sex Difference in Celiac Disease in Undiagnosed Populations: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2019 Sep;17(10):1954-1968.e13. doi: 10.1016/j.cgh.2018.11.013. Epub 2018 Nov 16. PMID 30448593
- [Result] Singh P, Arora A, Strand TA, Leffler DA, Catassi C, Green PH, Kelly CP, Ahuja V, Makharia GK. Global Prevalence of Celiac Disease: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2018 Jun;16(6):823-836.e2. doi: 10.1016/j.cgh.2017.06.037. Epub 2018 Mar 16. PMID 29551598
- [Result] Lindfors K, Ciacci C, Kurppa K, Lundin KEA, Makharia GK, Mearin ML, Murray JA, Verdu EF, Kaukinen K. Coeliac disease. Nat Rev Dis Primers. 2019 Jan 10;5(1):3. doi: 10.1038/s41572-018-0054-z. PMID 30631077
- [Result] Jansen M, van Zelm M, Groeneweg M, Jaddoe V, Dik W, Schreurs M, Hooijkaas H, Moll H, Escher J. The identification of celiac disease in asymptomatic children: the Generation R Study. J Gastroenterol. 2018 Mar;53(3):377-386. doi: 10.1007/s00535-017-1354-x. Epub 2017 Jun 6. PMID 28589338
- [Result] Csizmadia CG, Mearin ML, von Blomberg BM, Brand R, Verloove-Vanhorick SP. An iceberg of childhood coeliac disease in the Netherlands. Lancet. 1999 Mar 6;353(9155):813-4. doi: 10.1016/S0140-6736(99)00243-3. No abstract available. PMID 10459972
- [Result] Steens RF, Csizmadia CG, George EK, Ninaber MK, Hira Sing RA, Mearin ML. A national prospective study on childhood celiac disease in the Netherlands 1993-2000: an increasing recognition and a changing clinical picture. J Pediatr. 2005 Aug;147(2):239-43. doi: 10.1016/j.jpeds.2005.04.013. PMID 16126057
- [Result] Meijer CR, Schweizer JJ, Peeters A, Putter H, Mearin ML. Efficient implementation of the 'non-biopsy approach' for the diagnosis of childhood celiac disease in the Netherlands: a national prospective evaluation 2010-2013. Eur J Pediatr. 2021 Aug;180(8):2485-2492. doi: 10.1007/s00431-021-04068-1. Epub 2021 Apr 15. PMID 33856540
- [Result] Shamir R, Hernell O, Leshno M. Cost-effectiveness analysis of screening for celiac disease in the adult population. Med Decis Making. 2006 May-Jun;26(3):282-93. doi: 10.1177/0272989X06289012. PMID 16751327
- [Result] Wolters VM, Wijmenga C. Genetic background of celiac disease and its clinical implications. Am J Gastroenterol. 2008 Jan;103(1):190-5. doi: 10.1111/j.1572-0241.2007.01471.x. PMID 18184122
- [Result] Tran TM, Aghili A, Li S, Ongoiba A, Kayentao K, Doumbo S, Traore B, Crompton PD. A nested real-time PCR assay for the quantification of Plasmodium falciparum DNA extracted from dried blood spots. Malar J. 2014 Oct 4;13:393. doi: 10.1186/1475-2875-13-393. PMID 25282516
- [Result] McCabe ER. Utility of PCR for DNA analysis from dried blood spots on filter paper blotters. PCR Methods Appl. 1991 Nov;1(2):99-106. doi: 10.1101/gr.1.2.99. No abstract available. PMID 1842936
- [Result] Shaik M, Shivanna DK, Kamate M, Ab V, Tp KV. Single Lysis-Salting Out Method of Genomic DNA Extraction From Dried Blood Spots. J Clin Lab Anal. 2016 Nov;30(6):1009-1012. doi: 10.1002/jcla.21972. Epub 2016 Apr 13. PMID 27074880
- [Result] Karhus LL, Thuesen BH, Skaaby T, Rumessen JJ, Linneberg A. The distribution of HLA DQ2 and DQ8 haplotypes and their association with health indicators in a general Danish population. United European Gastroenterol J. 2018 Jul;6(6):866-878. doi: 10.1177/2050640618765506. Epub 2018 Mar 8. PMID 30023064
- [Result] Ruiz-Ortiz E, Montraveta M, Cabre E, Herrero-Mata MJ, Pujol-Borrell R, Palou E, Faner R. HLA-DQ2/DQ8 and HLA-DQB1*02 homozygosity typing by real-time polymerase chain reaction for the assessment of celiac disease genetic risk: evaluation of a Spanish celiac population. Tissue Antigens. 2014 Dec;84(6):545-53. doi: 10.1111/tan.12472. PMID 25413104
- [Result] Rouvroye MD, van Zijtveld S, Bonnet P, Spierings E, Bontkes HJ. HLA-DQ Typing Kits in Diagnosis and Screening for Celiac Disease. Genet Test Mol Biomarkers. 2019 Jun;23(6):418-422. doi: 10.1089/gtmb.2018.0329. Epub 2019 May 8. PMID 31066583
- [Result] Fasano ME, Dametto E, D'Alfonso S. HLA Genotyping: Methods for the Identification of the HLA-DQ2,-DQ8 Heterodimers Implicated in Celiac Disease (CD) Susceptibility. Methods Mol Biol. 2015;1326:79-92. doi: 10.1007/978-1-4939-2839-2_9. PMID 26498615
- [Result] Meijer CR, Auricchio R, Putter H, Castillejo G, Crespo P, Gyimesi J, Hartman C, Kolacek S, Koletzko S, Korponay-Szabo I, Ojinaga EM, Polanco I, Ribes-Koninckx C, Shamir R, Szajewska H, Troncone R, Villanacci V, Werkstetter K, Mearin ML. Prediction Models for Celiac Disease Development in Children From High-Risk Families: Data From the PreventCD Cohort. Gastroenterology. 2022 Aug;163(2):426-436. doi: 10.1053/j.gastro.2022.04.030. Epub 2022 Apr 26. PMID 35487291
- [Result] Wessels MM, Vriezinga SL, Koletzko S, Werkstetter K, Castillejo-De Villasante G, Shamir R, Hartman C, Putter H, van der Pal SM, Wijmenga C, Bravi E, Mearin ML; PreventCD Study Group. Impact on parents of HLA-DQ2/DQ8 genotyping in healthy children from coeliac families. Eur J Hum Genet. 2015 Mar;23(3):405-8. doi: 10.1038/ejhg.2014.113. Epub 2014 Jun 11. PMID 24916643
- [Result] Roy A, Pallai M, Lebwohl B, Taylor AK, Green PH. Attitudes Toward Genetic Testing for Celiac Disease. J Genet Couns. 2016 Apr;25(2):270-8. doi: 10.1007/s10897-015-9867-z. Epub 2015 Aug 2. PMID 26233331
- [Result] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226